CLINICAL TRIAL: NCT01144819
Title: Platelet Inhibition in the Acute Phase of ST-segment Elevation Myocardial Infarction
Brief Title: Platelet Inhibition in the Acute Phase of STEMI
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: AP Moeller Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 23374
Record Dates: First submitted 2010-03-26; First posted 2010-06-16 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Acute Myocardial Infarction; Antiplatelet Therapy; ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: STEMI; Acute myocardial infarction; Antiplatelet therapy; aspirin; clopidogrel; VerifyNow aggregometry; Multiplate aggregometry
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample 1:
  * Whole blood (Platelet aggregation tests and flowcytometry)
  * Serum
  * S-Thromboxane B2
  * S-Trombopoeitin
  * S-P-selectin
  * Plasma
  * DNA
  * RNA
  Blood sample 2:
  * Whole blood
  * Plasma
  Blood sample 3:
  * Whole blood
  * Plasma
  Blood sample 4:
  * Whole blood (Platelet aggregation tests and flowcytometry)
  * Serum
  * S-Thromboxane B2
  * S-Trombopoeitin
  * S-P-selectin
  * Plasma
  * DNA
  * RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI: Patients with STEMI according to ESC STEMI guidelines: Age above 18 years and able to give written, informed consent to participation in the project.

SUMMARY:
Background:

Dual antithrombotic treatment with aspirin and clopidogrel is recommended in patients with ST elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI). The European Society of Cardiology (ESC) Guidelines recommend a bolus dose of aspirin of 250-500 mg and a 600 mg bolus dose of clopidogrel as soon as STEMI is suspected. Studies have shown that more newly produced platelets are present in the acute phase of STEMI, and it is likely that these immature platelets are haemostatically more active and might be of importance in thrombus formation.

The enhanced platelet reactivity may reduce the effect of aspirin and clopidogrel in the acute phase of STEMI compared to measurements made in the same patients 3 months after primary PCI.

Aim:

This study aims to compare platelet response to aspirin and clopidogrel in the acute phase of STEMI with the platelet response in the same patients 3 months after STEMI .

Design:

This study is an observational follow-up study.

Materials and methods:

46 patients with STEMI referred to primary PCI at Aarhus University Hospital, Skejby will be included in the study. A total of 3 blood samples are obtained in the acute phase of STEMI: Prior to primary PCI (Blood sample 1), at 4 hours (Blood sample 2) and at 12 hours (Blood sample 3) after administration of loading dose aspirin and clopidogrel. When patients are in a stable phase 3 month later, a final blood sample is taken (Blood sample 4). The blood is analyzed 30 minutes after withdrawal of blood by the platelet aggregation test Multiplate® aggregometry (agonists: Collagen, arachidonic acid and adenosinediphosphate) and VerifyNow® arachidonic acid and P2Y12 aggregometry. Platelet count, volume and the immature platelet fraction (IPF) will be measured using Sysmex® flowcytometry.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Patients with ST-segment elevation myocardial infarction (STEMI) referred to primary PCI at University Hospital of Aarhus, Skejby.

Exclusion Criteria:

* Treatment with NSAID, ticlopidine and dipyramidole.
* Treatment with anticoagulants (Vitamin K antagonists)
* Patients diagnosed with platelet disease or haemophilia.
* Patients unable to give written, informed consent to participation in this project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of the Central Denmark Region.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Difference between aggregation induced by agonist collagen (1 μg/ml) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist collagen (1 μg/ml) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist collagen (1 μg/ml) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist arachidonic acid (1,0 mM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist arachidonic acid (1,0 mM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist arachidonic acid (1,0 mM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist adenosine diphosphate (6,4 µM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist adenosine diphosphate (6,4 µM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist adenosine diphosphate (6,4 µM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist adenosine diphosphate (20 µM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist adenosine diphosphate (20 µM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation induced by agonist adenosine diphosphate (20 µM) measured by Multiplate® Aggregometry (Unit=AUC). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation measured by VerifyNow® Aggregometry using the ASPI-kit (Unit = ARU). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation measured by VerifyNow® Aggregometry using the ASPI-kit (Unit = ARU). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation measured by VerifyNow® Aggregometry using the ASPI-kit (Unit = ARU). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation measured by VerifyNow® Aggregometry using the P2Y12-kit (Unit = PRU). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation measured by VerifyNow® Aggregometry using the P2Y12-kit (Unit = PRU). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference between aggregation measured by VerifyNow® Aggregometry using the P2Y12-kit (Unit = PRU). | Approximately 2-3 months
  Outcome is the difference between aggregation measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.

SECONDARY OUTCOMES:
Difference in immature platelet fraction measured by Sysmex® flowcytometry. | Approximately 2-3 months
  Outcome is the difference between measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after administration of LD aspirin and clopidogrel.
Difference in serum P-selectin | Approximately 2-3 months
  Outcome is the difference between measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after administration of LD aspirin and clopidogrel.
Difference in serum trombopoietin | Approximately 2-3 months
  Outcome is the difference between measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after administration of LD aspirin and clopidogrel.
Difference in serum thromboxane B2 | Approximately 2-3 months
  Outcome is the difference between measurements. In this case between:
  Blood sample 1: Obtained immediately before primary PCI in the catherization laboratory. The blood sample is obtained from the femoral artery catheter.
  Blood sample 4: 2-3 months after administration of LD aspirin and clopidogrel.
Difference in immature platelet fraction measured by Sysmex® flowcytometry. | Approximately 2-3 months
  Outcome is the difference between measurements. In this case between:
  Blood sample 2: 4 hours after administration of loading dose (LD) aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.
Difference in immature platelet fraction measured by Sysmex® flowcytometry. | Approximately 2-3 months
  Outcome is the difference between measurements. In this case between:
  Blood sample 3: 12 hours after administration of LD aspirin and clopidogrel.
  Blood sample 4: 2-3 months after primary PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Steen D Kristensen, MD, DMSc, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Central Jutland, Denmark

REFERENCES:
- [Result] Funck-Jensen KL, Dalsgaard J, Grove EL, Hvas AM, Kristensen SD. Increased platelet aggregation and turnover in the acute phase of ST-elevation myocardial infarction. Platelets. 2013;24(7):528-37. doi: 10.3109/09537104.2012.738838. Epub 2012 Dec 5. PMID 23216571